CLINICAL TRIAL: NCT06683612
Title: A Phase 1b, Open-label Study of PIPE-791 to Determine Brain and Lung Lysophosphatidic Acid Receptor 1 (LPA1) Occupancy, by [18F] PIPE-497 PET Imaging in Healthy Volunteers, Volunteers With Progressive Multiple Sclerosis, and Volunteers With Idiopathic Pulmonary Fibrosis
Brief Title: PET Study of PIPE-791 in Healthy Volunteers and Volunteers With PrMS and IPF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Contineum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTX-791-102
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF); Idiopathic Pulmonary Fibrosis; Multiple Sclerosis; Multiple Sclerosis, MS; Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Progressive; Multiple Sclerosis, Secondary Progressive; Healthy; Healthy Volunteers
Keywords: remyelination; MS; multiple sclerosis; PrMS; PPMS; SPMS; primary progressive MS; primary progressive multiple sclerosis; secondary progressive multiple sclerosis; secondary progressive MS; LPA1; PMS; idiopathic pulmonary fibrosis; IPF; neuroinflammation; PIPE-791; demyelinating diseases; autoimmune diseases; pathologic processes; demyelinating autoimmune diseases, CNS; autoimmune diseases of the nervous system; nervous system diseases; immune diseases; sclerosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive; Neuroinflammatory Diseases; Demyelinating Diseases; Autoimmune Diseases; Pathologic Processes; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Immune System Diseases; Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy volunteers, brain PET imaging (Experimental)
  Interventions: Drug: PIPE-791
- Healthy volunteers, lung PET imaging (Experimental)
  Interventions: Drug: PIPE-791
- Volunteers with PrMS (Experimental)
  Interventions: Drug: PIPE-791
- Volunteers with IPF (Experimental)
  Interventions: Drug: PIPE-791

INTERVENTIONS:
Drug: PIPE-791 — Subjects will receive a single oral dose of PIPE-791.

SUMMARY:
This is a study of PIPE-791, an investigational study drug to treat progressive multiple sclerosis (MS) and idiopathic pulmonary fibrosis (IPF). The purpose of this study is to find out how much of the study drug gets into the brain and lung, and what the side effects and blood levels of the study drug are in healthy volunteers and patients.

Participants will:

* Take a single dose of the study drug
* Give many samples of blood and urine
* Have multiple PET scans

ELIGIBILITY:
Main Inclusion Criteria

* All parts: male volunteers or female volunteers of non-childbearing potential; agree to follow the contraception requirements of the trial, and able to give fully informed written consent.
* Part A: normotensive volunteers, deemed healthy on the basis of a clinical history, medical examinations, ECG, vital signs, and laboratory tests of blood and urine.
* Part B: volunteers with a diagnosis of PPMS or SPMS by a neurologist, according to the 2017 Revised McDonald Criteria.
* Part C: volunteers with a diagnosis of IPF by a pulmonologist, according to the 2018 American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Society (ALAT) Clinical Practice Guideline, within 7 years before screening.

Main Exclusion Criteria

* Positive tests for hepatitis B and C, human immunodeficiency virus (HIV)
* Severe adverse reaction to any drug; sensitivity to trial medication
* Drug or alcohol abuse
* Smoking or use of tobacco or nicotine-containing products from 7 days before screening, until the final visit
* Use of a prescription medicine (except hormone replacement therapy [HRT] in women, and medications for participants with PrMS and IPF at the discretion of the investigator), or any substance known to interact with cytochrome p450 (CYP)3A enzymes (including St. John's wort and foodstuffs such as grapefruit juice) during the 28 days before the first dose of PIPE-791
* Use of any other over-the-counter medicine, with the exception of acetaminophen (paracetamol) during the 7 days before the first dose of PIPE-791, or received vaccine against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), during the 7 days before screening
* Participation in other clinical trials of unlicensed medicines, or loss of more than 400 mL blood, within the 3 months before the baseline PET scan
* Vital signs or ECGs outside the acceptable range at screening
* Clinically relevant abnormal findings at the screening assessments, including C-SSRS and MRI (Parts A [brain PET imaging arm] and B only)
* Acute or chronic illness (except PrMS and IPF in Parts B and C, respectively)
* Clinically relevant abnormal medical history or concurrent medical condition
* Possibility that volunteer will not cooperate
* Contraindications to MRI (Parts A [brain PET imaging arm] and B only), computed tomography (CT), PET, or arterial cannulation procedures
* Significant exposure to research-related radiation or other radiation exposure (exceeding 10 mSv when added to exposure from this study) within the previous 12 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
LPA1 occupancy as determined by regional total volume of distribution (VT) at each brain scan. | Baseline to up to 28 days post-dose
LPA1 occupancy as determined by regional total volume of distribution (VT) at each lung scan. | Baseline to up to 28 days post-dose

SECONDARY OUTCOMES:
The relationship between PIPE-791 plasma concentration and brain and lung LPA1 occupancy. | Baseline to up to 28 days post-dose
The PIPE-791 EC50 (i.e., the plasma concentration of PIPE-791 associated with 50% occupancy of LPA1) in the brain and lungs. | Baseline to up to 28 days post-dose
Pharmacokinetics (PK): blood concentration levels of PIPE-791 | Baseline to up to 28 days post-dose
Safety and tolerability: Treatment-Emergent Adverse Events (TEAE) | Baseline to up to 32 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, MD, Study Director — Contineum Therapeutics
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No